CLINICAL TRIAL: NCT06621628
Title: Polarized Light Therapy and Hand Grip Strengthening Exercises in Patients With CREST Syndrome.
Brief Title: Polarized Light Therapy in Patients With CREST Syndrome.
Acronym: CREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Ismailia National University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Moeim Abo EL Ros, Lecturer of Physical Therapy for Pediatrics and its Surgeries, New Ismailia National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004063
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: CREST Syndrome
Keywords: Polarized light therapy; Resisted exercise; CREST syndrome; Modified Rodnon skin score; and Hand Grip Dynamometer
MeSH Terms: conditions — CREST Syndrome

STUDY DESIGN:
Intervention Model Description: to evaluate the efficacy of the Polarized light therapy and Hand Grip Strengthening exercises in patients with CREST syndrome.
Who Masked: Participant
Masking Description: masking was done by sealed envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Study group A (Experimental): This group included 20 patients who had CREST syndrome with scleroderma in the dorsum of hands and who received the BLT with traditional physical therapy program (stretching, strengthening and active exercise) patients received 3 sessions per week for 12 weeks (3 months),time of session is 15 minutes.
  Interventions: Other: stretching, strengthening exercises and active exercises
- study group B (Experimental): This group included 20 patients who have CREST syndrome with scleroderma in the dorsum of hands and who received resisted exercise with traditional physical therapy program (stretching, strengthening and active exercise) patients received 3 sessions per week for 12 weeks (3 months), time of session is 15 minutes
  Interventions: Other: stretching, strengthening exercises and active exercises
- study group C (Experimental): This group included 20 patients who had CREST syndrome with scleroderma in the dorsum of hands and who received combination of (bipotron light therapy and resisted exercise) with traditional physical therapy program (stretching, strengthening and active exercise) exercise program (stretching, strengthening and active exercise).patients received 3 sessions per week for 12weeks (3 months), time of session is 15 minutes
  Interventions: Other: stretching, strengthening exercises and active exercises

INTERVENTIONS:
Other: stretching, strengthening exercises and active exercises — Bioptron light therapy device, resisted exercises and stretching exercises
  Other Names: resisted exercise, stretching and active exercises

SUMMARY:
to evaluate the efficacy of the Polarized light therapy and Hand Grip Strengthening exercises in patients with CREST syndrome

DETAILED DESCRIPTION:
Measurement of the skin thickness via the modified Rodnon skin score (RSS) and Hand Grip Dynamometer (HGD) . Methods:- Sixty patients, who had hand involvement of patients with CREST syndrome, were participated in the study. Their ages were ranged from 16 to 45 years. The participants were selected from the dermatology departments of Cairo university hospitals and Om El-Misrieen hospital, randomly distributed into three equal groups. Group A: (Study group): This group included 20 patients who had CREST syndrome with scleroderma in the dorsum of hands and who received the BLT with traditional physical therapy program (stretching, strengthening and active exercise) patients received 3 sessions per week for 12 weeks (3 months),time of session is 15 minutes. Group B: This group included 20 patients who have CREST syndrome with scleroderma in the dorsum of hands and who received resisted exercise with traditional physical therapy program (stretching, strengthening and active exercise) patients received 3 sessions per week for 12 weeks (3 months), time of session is 15 minutes and Group C:This group included 20 patients who had CREST syndrome with scleroderma in the dorsum of hands and who received combination of (BLT and resisted exercise) with traditional physical therapy program (stretching, strengthening and active exercise) exercise program (stretching, strengthening and active exercise).patients received 3 sessions per week for 12weeks (3 months), time of session was 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The patients' ages ranged from 16 to 21 years.
* Patients who had hand involvement of patients with CREST syndrome particularly dorsum of the hand.
* All patients were conscious.
* All patients were randomly chosen (male and female).

Exclusion Criteria:

* Patients who are diabetic or hypertensive.
* Patients those familiar with the BLT and resisted exercise via the hand grip strengthener.
* Patients with hemorrhage specially hemorrhage of digestive system and those with bleeding per rectum.
* Patients with severe fungal diseases and acute viral diseases.
* Patients with active tuberculosis and tumors as well as those with peacemakers.
* Patients with polyneuropathy.
* Patients with thyroid problems

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
skin thickness | 12 weeks
  modified random skin score
hand grip strength and pinch gauge | 12 weeks
  Hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Zakaria E Mowafy, Ph.D, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Khadra Mohamed Ali, Ismailia
  - Mohamed Abdel Moenem Abo El Ros, Ismailia

IPD SHARING:
Plan to Share IPD: No
this proposal was assigned to evaluate skin thickness and pinch gauge concerning hand function using Bioptron light therapy in patients with crest syndrome

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT06621628/Prot_SAP_ICF_000.pdf